CLINICAL TRIAL: NCT02898480
Title: Changes in the Diameter of Retinal Vessels After Remote Ischemic Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RIK-DVA
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2017-11

CONDITIONS: Retinal Artery Occlusion; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Artery Occlusion; Retinal Vein Occlusion

ARMS (1):
- Remote ischemic conditioning (Experimental)
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Briefly reversible restricting of blood flow to upper limb in four cycles of 5 minutes of inflation at 200mm Hg followed by 5 minutes of deflation.

SUMMARY:
Remote ischemic conditioning (RIC) is a therapeutic strategy for protecting organs or tissue against the detrimental effects of acute ischemia-reperfusion injury. It remains unknown whether this can be used in retinal vascular occlusive diseases. The purpose of the present study is to examine whether the autoregulation of retinal vessel diameters in normal persons change after remote ischemic conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Normal persons

Exclusion Criteria:

* Present or previous eye disease
* Use of medications except anti-conceptive
* Epilepsy
* Pregnancy or lactation

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11-14 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Diameter change of retinal vessel | immediate